CLINICAL TRIAL: NCT01077024
Title: Smoking-Cessation and Stimulant Treatment (S-CAST): Evaluation of the Impact of Concurrent Outpatient Smoking-Cessation and Stimulant Treatment on Stimulant-Dependence Outcomes
Brief Title: Smoking-Cessation and Stimulant Treatment (S-CAST)
Acronym: S-CAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theresa Winhusen, Professor; Director, Center for Addiction Research, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0046; 5U10DA013732 (NIH); 3U10DA013732-10 (NIH)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cocaine Dependence; Methamphetamine Dependence; Nicotine Dependence
Keywords: Stimulant treatment; Smoking Cessation
MeSH Terms: conditions — Cocaine-Related Disorders; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoking-cessation treatment + substance treatment as usual (Experimental)
  Interventions: Other: Smoking-cessation treatment
- Substance-treatment as usual (No Intervention): Treatment as usual is outpatient stimulant-dependence treatment as typically provided by the participating site.

INTERVENTIONS:
Other: Smoking-cessation treatment — Smoking cessation treatment includes four components: 1. brief weekly individual smoking-cessation counseling study weeks 1-10; 2. extended-release (XL) bupropion (300 mg/day)study weeks 1-10; 3. nicotine inhaler (6-16 cartridges per day ad libitum)during the post-quit treatment phase; 4. prize-based contingency management during the post-quit treatment phase.
  Arms: Smoking-cessation treatment + substance treatment as usual

SUMMARY:
The primary objective of this study is to evaluate the impact of substance-abuse treatment as usual plus smoking-cessation treatment (TAU+SCT), relative to substance-abuse treatment as usual (TAU), on drug-abuse outcomes. Specifically, this study will evaluate whether concurrent smoking-cessation treatment improves, worsens, or has no effect on stimulant-use outcomes in smokers who are in outpatient substance-abuse treatment for cocaine or methamphetamine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cocaine/methamphetamine dependence
* Smoked cigarettes for at least 3 months
* Currently smoking > 6 cigarettes/day
* Have an interest in quitting smoking
* Enrolled in outpatient treatment at a participating site

Exclusion Criteria:

* Clinical diagnosis of current alcohol or sedative dependence, bipolar disorder; or a life-time diagnosis of anorexia nervosa or bulimia
* Seeking/receiving treatment for opiate-agonist replacement therapy
* Medical conditions that could compromise participant safety
* Taking medications with known/potential interactions with bupropion
* Hypersensitivity to bupropion, nicotine, or menthol
* Pregnant or breastfeeding
* Abnormal ECG
* Recent smoking cessation treatment
* Use of tobacco products other than cigarettes in the past week
* Likely to enter residential/inpatient treatment within 10 weeks
* Have all stimulant-positive urine drug screens during screening/baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, Ph.D., Principal Investigator — University of Cincinnati
Locations (12):
- United States (12):
  - La Frontera, Tucson, Arizona
  - Matrix Institute on Addictions, Rancho Cucamonga, California
  - Tarzana Treatment Centers, Tarzana, California
  - Gateway, Jacksonville, Florida
  - Gibson Recovery Center, Inc., Cape Girardeau, Missouri
  - Maryhaven, Columbus, Ohio
  - ADAPT, Roseburg, Oregon
  - Addiction Medicine Services, Pittsburgh, Pennsylvania
  - Lexington/Richland Alcohol and Drug Abuse Council, Columbia, South Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina
  - Dorchester, Summerville, South Carolina
  - Nexus Recovery Center, Dallas, Texas

REFERENCES:
- [Derived] Winhusen TM, Theobald J, Lewis DF. Substance use outcomes in cocaine-dependent tobacco smokers: A mediation analysis exploring the role of sleep disturbance, craving, anxiety, and depression. J Subst Abuse Treat. 2019 Jan;96:53-57. doi: 10.1016/j.jsat.2018.10.011. Epub 2018 Oct 26. PMID 30466549
- [Derived] Winhusen TM, Brigham GS, Kropp F, Lindblad R, Gardin JG 2nd, Penn P, Hodgkins C, Kelly TM, Douaihy A, McCann M, Love LD, DeGravelles E, Bachrach K, Sonne SC, Hiott B, Haynes L, Sharma G, Lewis DF, VanVeldhuisen P, Theobald J, Ghitza U. A randomized trial of concurrent smoking-cessation and substance use disorder treatment in stimulant-dependent smokers. J Clin Psychiatry. 2014 Apr;75(4):336-43. doi: 10.4088/JCP.13m08449. PMID 24345356
- [Derived] Winhusen TM, Kropp F, Theobald J, Lewis DF. Achieving smoking abstinence is associated with decreased cocaine use in cocaine-dependent patients receiving smoking-cessation treatment. Drug Alcohol Depend. 2014 Jan 1;134:391-395. doi: 10.1016/j.drugalcdep.2013.09.019. Epub 2013 Sep 27. PMID 24128381
- [Derived] Winhusen TM, Adinoff B, Lewis DF, Brigham GS, Gardin JG 2nd, Sonne SC, Theobald J, Ghitza U. A tale of two stimulants: mentholated cigarettes may play a role in cocaine, but not methamphetamine, dependence. Drug Alcohol Depend. 2013 Dec 15;133(3):845-51. doi: 10.1016/j.drugalcdep.2013.09.002. Epub 2013 Sep 11. PMID 24075226
- See also: NIDA Clinical Trials Network — http://www.drugabuse.gov/CTN/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Started | 267 | 271
Completed | 236 | 243
Not Completed | 31 | 28
Not completed — Lost to Follow-up | 20 | 14
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Incarcerated | 7 | 8
Not completed — Other | 4 | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis was performed on the Intent-to-Treat population, which was the population of randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual | Total
Number analyzed (Participants) | 267 | 271 | 538
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 266 | 271 | 537
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 136 | 258
  Male | 145 | 135 | 280
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 83 | 88 | 171
  White | 162 | 158 | 320
  More than one race | 4 | 13 | 17
  Unknown or Not Reported | 14 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 33 | 67
  Not Hispanic or Latino | 230 | 236 | 466
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 267 | 271 | 538
Weight [Mean (Standard Deviation); unit: pounds] | 184.8 (43.77) | 183.3 (44.21) | 184.0 (43.96)

OUTCOME MEASURES:

1. Primary Outcome: Stimulant-free Weeks Assessed by Self-report and Twice-weekly Urine Drug Screens
Description: Stimulant-free week results (no cocaine, methamphetamine and amphetamine use) were obtained by combining the urine drug screens (UDS) and the self-reported Timeline Follow-Back (TLFB). At the group level, this outcome translates into the percentage of weeks in each study arm that are stimulant-free.
Time Frame: Week 16
Measure: Number; unit: percentage of weeks
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 267 | 271
percentage of weeks | 77.7 [0.6940 to 1.3196] | 78.0 [0.6940 to 1.3196]

2. Secondary Outcome: Point-prevalence Abstinence (Smoking Outcome)
Description: point-prevalence abstinence defined as not smoking in the previous seven days based on self-report and confirmed with a Carbon Monoxide (CO) level ≤ 8 ppm
Time Frame: Week 10 assessment
Measure: Number; unit: percentage of participants
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 267 | 271
percentage of participants | 25.5 | 2.2

3. Secondary Outcome: Four Week Continuous Smoking Abstinence
Description: A combination of daily self-reported smoking data and weekly carbon monoxide levels were used to determine continuous abstinence during post-quit days 15 - 42.
Time Frame: Post-quit days 15-42
Measure: Number; unit: percentage of participants
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 267 | 271
percentage of participants | 6.7 | 0.0

4. Secondary Outcome: Stimulant-free Results at 3-month Visit
Description: At the 3-month follow-up visit, percentage of participants with a negative urine drug screen for stimulant use and no stimulant use days reported during the past 28 days based on Timeline Follow-back.
Time Frame: 3-month follow-up visit
Population: This outcome was only compared for participants who attended the 3-month follow-up visit (n=226 and n=240, respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 226 | 240
percentage of participants | 74.3 | 68.8

5. Secondary Outcome: Point-prevalence Abstinence (Smoking Outcome) 3 Month Visit
Description: as for outcome 2
Time Frame: 3- month follow-up visits
Measure: Number; unit: percentage of participants
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 267 | 271
percentage of participants | 19.1 | 3.0

6. Secondary Outcome: Stimulant-free Results at 6-month Visit
Description: At the 6-month follow-up visit, percentage of participants with a negative urine drug screen for stimulant use and no stimulant use days reported during the past 28 days based on Timeline Follow-back.
Time Frame: 6 - months follow-up visit
Population: This outcome was only compared for participants who attended the 6-month follow-up visit (n=210 and n=218, respectively).
Measure: Number; unit: percentage of participants
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 210 | 218
percentage of participants | 69.5 | 71.6

7. Secondary Outcome: Point-prevalence Abstinence (Smoking Outcome) 6 Month Visit
Description: as for outcome 2
Time Frame: 6 month visit
Measure: Number; unit: percentage of participants
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Number analyzed (Participants) | 267 | 271
percentage of participants | 13.1 | 3.7

ADVERSE EVENTS:
Time Frame: A systematic collection of adverse events occurred from the time of consent to the 10th week final visit. Serious adverse events discovered unsystematically were collected through 30 days following the 10th week final visit.
Description: Investigators systematically interviewed participants at each study week regarding any untoward events occurring since the last study visit.
Arm/Group | Smoking-cessation Treatment + Substance Treatment as Usual | Substance-treatment as Usual
Serious Adverse Events (participants affected / at risk) | 14/267 | 9/271
Other Adverse Events (participants affected / at risk) | 181/267 | 89/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoking-cessation Treatment + Substance Treatment as Usual (N=267) | Substance-treatment as Usual (N=271)
Angina Pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constiipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) — Death of unknown cause
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoking-cessation Treatment + Substance Treatment as Usual (N=267) | Substance-treatment as Usual (N=271)
Dry mouth (Gastrointestinal disorders) | 14 (14) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (18) | 7 (7)
Toothache (Gastrointestinal disorders) | 14 (14) | 15 (15)
Nasopharyngitis (Infections and infestations) | 19 (19) | 19 (19)
Sinusitis (Infections and infestations) | 9 (9) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 13 (13)
Headache (Nervous system disorders) | 34 (34) | 13 (13)
Anxiety (Psychiatric disorders) | 20 (20) | 5 (5)
Insomnia (Psychiatric disorders) | 21 (21) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 0 (0)

LIMITATIONS AND CAVEATS:
Stimulant use was relatively low throughout the study; this may have limited our ability to make inferences about the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No